CLINICAL TRIAL: NCT07064525
Title: A Multi-center, Randomized, Double-blind, Parallel, Phase 2b Study to Evaluate the Efficacy and Safety of SPC1001 Low in Patients With Essential Hypertension
Brief Title: Evaluate the Efficacy and Safety of SPC1001 Low in Patients With Essential Hypertension
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-CAP-HTN-203
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hypertension (HTN); NYHA Class III Heart Failure; NYHA Class IV Heart Failure; Diabete Mellitus
Keywords: blood pressure; phase 2b; low dose combination therapy; candesartan; amlodipine; indapamide
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — SPC 5002

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SPC1001 Low (Active Comparator): low-dose combination therapy
  Interventions: Drug: SPC1001 Low
- SPC5002 (Active Comparator): low-dose combination therapy
  Interventions: Drug: SPC1001 Low; Drug: SPC5002
- SPC5003 (Active Comparator): low-dose combination therapy
  Interventions: Drug: SPC1001 Low; Drug: SPC5003
- SPC5004 (Active Comparator): low-dose combination therapy
  Interventions: Drug: SPC1001 Low; Drug: SPC5004

INTERVENTIONS:
Drug: SPC1001 Low — low-dose combination therapy
Drug: SPC5002 — low-dose combination therapy
  Arms: SPC5002
Drug: SPC5003 — low-dose combination therapy
  Arms: SPC5003
Drug: SPC5004 — low-dose combination therapy
  Arms: SPC5004

SUMMARY:
- Objective: This study aims to evaluate the safety and efficacy of the fixed-dose triple combination therapy (SPC1001 Low) of candesartan, amlodipine, and indapamide in adult patients with essential hypertension compared to dual-component therapies of each ingredient for 8 weeks. Additionally, it seeks to confirm the contribution of each component at low doses.

- Inclusion Criteria: Men and women aged 19 to 75 years whose blood pressure measured at the screening visit meets the following criteria.

- Exclusion Criteria: Patients whose blood pressure measured at the screening and randomization visits meets the criteria of MSSBP ≥180 mmHg or MSDBP ≥110 mmHg, among other conditions.

- Methods: This study is a multicenter, randomized, double-blind, parallel-group, phase 2b clinical trial to evaluate the safety and efficacy of the investigational drug after 8 weeks of administration.

Screening assessments will be conducted within 4 weeks prior to randomization, and patients who meet the inclusion and exclusion criteria at the screening visit will be enrolled in the study after providing informed consent. These participants will undergo a 2-week run-in period during which they will take a placebo and participate in a lifestyle modification program.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 19 to 75 years whose blood pressure measured at the screening visit meets the following criteria.

Exclusion Criteria:

* Patients whose blood pressure measured at the screening and randomization visits meets the criteria of MSSBP ≥180 mmHg or MSDBP ≥110 mmHg, among other conditions.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was determined by evaluating how mean sitting systolic blood pressure varied between the baseline measurement and week 8 | change in MSSBP from baseline at week 8

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Gangnam Medical Center, CHA University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
It is planned to be publicly available in the form of a future journal submission
Supporting Information: Study Protocol